CLINICAL TRIAL: NCT05446792
Title: Comparison Between Pelvic Floor Muscle Training and Pilates Exercises on Urinary Incontinence in Postmenopausal Women: Randomized Controlled Trial
Brief Title: Comparison Between Pelvic Muscle Training and Pilates Exercises for UI in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Laís Campos de Oliveira, Doctor Teacher Laís Campos de Oliveira, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMAP X Pilates in the UI
Record Dates: First submitted 2022-06-24; First posted 2022-07-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Urinary Incontinence
Keywords: Post-menopause; Pilates; Muscle training of pelvic floor
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The interventions will last for twelve weeks, three times a week, for one hour, on non days consecutive.
  The Pilates exercises group will perform stretching and strengthening exercises in a single series of 10 repetitions, totaling 10 exercises aimed at the main muscle groups.
  The Pelvic floor muscle training group will consist of 10 maximal voluntary contractions that must be maintained for at least 6 seconds (participants will be encouraged to sustain the maximal contraction for a longer time each week). The interval time between contractions will be the same seconds as the contraction. Participants will perform 4 sets of 10 contractions, and at the end of each set of 10 contractions, five fast contractions will be performed. Each series will be performed in one position: 1st lying in lateral decubitus, 2nd sitting, 3rd on all fours and 4th standing.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization of the sample will be confidential. A professional in the field who is unaware of the study and the participants will perform the draw through random numbers that will distribute the participants into two groups: Pelvic Floor Muscle Training Group (TMAP) (n= 20) and Pilates Exercise Group (PE) (n= 20). This same professional will deliver the answers in opaque envelopes, which will be sealed and contain the answer. Participants will be duly informed that they can be allocated to either of the two groups at the time of recruitment and selection and, in addition, the participants and the responsible researchers will know in which group each woman will participate at the time of delivery of the envelopes.
  The evaluations will be carried out before and after three months of interventions, by the same professionals, experienced in these evaluations, who will be blind to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle training (PFMT) (Active Comparator): For the intervention of the PFMT group, which is non-invasive, a physical therapist experienced in this type of training will carry out the sessions, which will be individualized, in a specific room for care ocused on pelvic physiotherapy, with a stretcher, air conditioning and a lock on the door, for the patient to feel safe.
  Interventions: Other: PFMT
- Pilates exercises (PE) (Experimental): For the intervention of the PE group, in the first week the protocol will be used to familiarize the participants with the exercises, where the correct execution of the movements will be demonstrated and each principle of the method will be explained: concentration, centralization, precision, breathing, control and fluidity; and for familiarization with the correct voluntary contraction of the PFM. Participants in the PE group will be instructed and reminded to voluntarily contract the PFM during each repetition of the Pilates strengthening exercises. During the stretching exercises, the participant will be instructed not to perform the contraction. The springs will be changed according to the evolution of the participants, by replacing them with a spring of greater resistance. Basic equipment such as: Cadillac Trapezio, Combo Chair, Universal Reformer, Ladder Barrel and Wall Unit will be used.
  Interventions: Other: PE

INTERVENTIONS:
Other: PFMT — The PFMT will consist of 10 maximum voluntary contractions that must be maintained for at least 6 seconds. Participants will be encouraged to sustain the maximum contraction for a longer time each week. The interval time between contractions will be the same seconds as the contraction. Participants will perform 4 sets of 10 contractions, and at the end of each set of 10 contractions, five fast contractions will be performed. Each series will be performed in one position: lying in lateral decubitus; seated; on all fours and standing.
  Arms: Pelvic floor muscle training (PFMT)
Other: PE — The PE group will be instructed and reminded to voluntarily contract the PFMs during each repetition of the Pilates strengthening exercises. During the stretching exercises, the participant will be instructed not to perform the contraction.
  The stretching and strengthening exercises will be performed in a single series of 10 repetitions, totaling 10 exercises aimed at the main muscle groups.
  Arms: Pilates exercises (PE)

SUMMARY:
Introduction: Urinary incontinence (UI) is a condition that affects around 40% of postmenopausal women and is therefore considered a public health problem. Conservative treatment is recommended, and pelvic floor muscle training (PMT) is considered the gold standard for this type of condition. However, other possibilities of exercises have been studied to achieve continence, such as Pilates exercises, which focus on the stabilizing muscles and request a voluntary contraction of the muscles of the pelvic floor (PFM), it is believed that it can recruit fibers from these muscles, improving muscle function and episodes of urinary incontinence. However, the literature is still inconclusive regarding the effects of Pilates exercises on urinary incontinence and PFM function. Objective: To compare the effects of 3 months of muscle training, through TMAP and Pilates exercises on the improvement of UI in postmenopausal women. Methods: 40 postmenopausal women with urinary incontinence will be randomly assigned to two intervention groups: pelvic floor muscle training and Pilates exercises. The evaluations will be carried out before the interventions and after three months of them, and will involve the following instruments: urinary incontinence and aspects related to quality of life, assessed using the International Consultation of Urinary Incontinence questionnaire Short Form (ICIQ-UI-SF); 7-day voiding diary, used to identify possible modifiable factors related to urination and its frequency; Pad-test used to identify and quantify UI; Feeling Scale, to portray the affective valence of the exercises; Female Sexual Function Index, which will assess female sexual function; Manometric assessment of muscle strength and PFM endurance with Epi-no; and Manometric evaluation by bidigital palpation using the PERFECT test. Shapiro Wilk tests will be performed to verify normality, Student's t or Mann Whitney U test according to parametric or non-parametric distribution, ANCOVA for comparison between groups in the post-intervention, considering the 95% confidence interval (p<0.05) . The data will be processed in the SPSS 25.0 program.

DETAILED DESCRIPTION:
The sample will be composed of 40 women in the post-menopausal period, that is, who are at least one year without menstruating, and who are aged between 50 and 70 years. The sample size calculation for this study was performed using the Bioestat 5.3 program (Mamirauá Institute, Amazonas, Brazil), taking into account the values of the ICIQ_SF instrument (name in English), made available in a previous study (SCHRADER et al., 2017). In this case, the post-intervention mean and standard deviation between the Pilates group (1.0 ± 1.15) and TMAP (3.42 ± 3.4) were used, with test power at 80% and alpha value at 0.05, which generated the need for 17 participants in each group. In order to meet eventual sample losses, 15% of participants will be added in each group, thus totaling 20 women in the Pilates group and 20 in the TMAP group.

The descriptive analysis of the data will be expressed in the form of mean, standard deviation and percentage delta of the difference. The verification of normality will occur by the Shapiro Wilk test. To verify if there are differences between the groups regarding the initial characteristics (age, weight, height and BMI), at the pre-intervention moment, the Student's t test will be used for independent samples or the Mann Whitney U test, in case the data show parametric or nonparametric distribution, respectively. For comparison between groups in the post-intervention ANCOVA will be used, with baseline data being used as covariates. If the data present a non-parametric characteristic, the comparison between the groups will be made using the Mann-Whitney U test, considering the difference between pre and post-intervention. The admitted confidence interval will be 95% (p<0.05). The data will be processed in the SPSS 25.0 program. Effect sizes (Cohen's d) will be calculated and considered small (0.20), medium (0.50) or large (0.80). For effect size calculations, the program GPower 3.1 (Franz Faul, Universitat Kiel, Germany) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Being naturally post-menopause (at least one year without menstruating);
* Demonstrate independence to carry out activities of daily living;
* Have a report of urinary loss when performing physical exertion.

Exclusion Criteria:

* Women who have had hysterectomy or oophorectomy surgery;
* Women who underwent cancer treatment with hormone therapy;
* Present cognitive deficits or neurological diseases;
* Practice any type of physical activity regularly in the last six months;
* Present inability to hire PFM (Oxford Scale < 1);
* Report pain or discomfort in the vulva or vagina;
* Present dyspareunia, vaginismus or pelvic organ prolapse greater than grade II in the Baden-Walker classification;
* Present symptoms of urinary infection at the time of evaluation;
* Have participated in previous pelvic floor reeducation programs.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
International Consultation of Urinary questionnaire Incontinence Short Form (ICIQ-UI-SF) | 3 months
  Specific quality of life questionnaire for each aspect related to UI. It consists of four questions; the sum of the first three questions gives the score, and the fourth describes the type of UI. The maximum total score is 21, and the higher the score, the worse the UI severity and disorder.
Pad-test | 3 months
  Identifies and quantifies UI. The participant will be instructed to empty the bladder and ingest 500 ml of water, then place a previously weighed absorbent. The participant performs provocative maneuvers that will increase intra-abdominal pressure such as coughing, jumping and crouching, lasting approximately one hour. Soon after, the absorbent will be weighed again. If the absorbent weight is greater than 2 grams, the result was positive, identifying the UI. The greater the final weight of the pad, the greater the amount of urinary loss.
Voiding diary | 3 months
  Identifies the frequency of urinary leakage. The participant will record, over the course of 7 days, at home, the number of episodes of urinary leakage during some effort, such as coughing, sneezing or jumping. If there are more than 3 urinary losses within a 7-day interval, the test is positive for UI.
Manometric assessment of muscle strength and PFM endurance | 3 months
  The manometer probe will be inserted and inflated in the participant's vaginal canal, until the participant feels the probe contacting the vaginal wall. The participant will be guided to contract the MAP. When the musculature contracts, an increase in pressure is observed on the device's display. You will be asked for three maximum contractions with 30 second rest intervals between contractions. The values will be recorded in mmHg and the duration of the contraction will be recorded in seconds. The higher the score, the stronger the MAPs are.
PERFECT test | 3 months
  As a complement to the manometric evaluation, bidigital palpation will be performed. The PFM strength and resistance level will be classified using the modified Oxford scale, where 0 is the absence of muscle strength and 5 means a strong contraction with movement correct "squeeze" and "suction". Participants will attempt maximum contractions in terms of strength and endurance three times, with 30-second rest intervals between contractions. The closer to a score of 5, the better the MAP.

SECONDARY OUTCOMES:
FSFI Questionnaire (Female Sexual Function Index) | 3 months
  To assess women's sexual function, the domains: desire, arousal, lubrication, orgasm, satisfaction and pain are used. It has 19 items. Each question presents a possibility of response with a pattern from 0 to 5, where at the end you can have the result of the scores of each domain and also of the total score, where values below or equal to 26.55 indicate sexual dysfunction.
Feeling Scale - Pleasure and displeasure during exercise | 3 months
  The affective valence scale will be used to measure the participants' feelings of pleasure/affection in relation to the exercises. The score goes from +5 meaning pleasure during the exercise with a feeling of "very good"; down to -5, meaning displeasure, presenting the feeling of "very bad" during the execution of the exercise. The closer to +5, the more pleasure in performing the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Laís C Oliveira, PhD, Principal Investigator — Universidade Estadual do Norte do Paraná; Raphael G Oliveira, PhD, Study Chair — Universidade Estadual do Norte do Paraná
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Andrade RL, Bo K, Antonio FI, Driusso P, Mateus-Vasconcelos ECL, Ramos S, Julio MP, Ferreira CHJ. An education program about pelvic floor muscles improved women's knowledge but not pelvic floor muscle function, urinary incontinence or sexual function: a randomised trial. J Physiother. 2018 Apr;64(2):91-96. doi: 10.1016/j.jphys.2018.02.010. Epub 2018 Mar 21. PMID 29574170
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- Available data/document: Approval of the Ethics Committee for Research with Human Beings in Brazil — https://plataformabrasil.saude.gov.br/login.jsf